CLINICAL TRIAL: NCT01985750
Title: Understanding the Importance of Plasticity in the Brain Mechanisms of Dyspnoea Perception
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OX-KP001
Record Dates: First submitted 2013-10-29; First posted 2013-11-15 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyspnea; fmri; d-cycloserine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: d-cycloserine or placebo (Placebo Comparator): Other Names:
  comparison of d-cycloserine or placebo on enhancing the beneficial effects of pulmonary rehabilitation on breathlessness perception
  250mg d-cycloserine or identical placebo given immediately to the first 4 sessions of a 6-week course pulmonary rehabilitation
  Interventions: Drug: placebo
- D-cycloserine (Active Comparator): Placebo Comparator: Drug: d-cycloserine or placebo
  Other Names:
  comparison of d-cycloserine or placebo on enhancing the beneficial effects of pulmonary rehabilitation on breathlessness perception
  250mg d-cycloserine or identical placebo given immediately to the first 4 sessions of a 6-week course pulmonary rehabilitation
  Interventions: Drug: d-cycloserine

INTERVENTIONS:
Drug: d-cycloserine — 250mg d-cycloserine or identical placebo given immediately to the first 4 sessions of a 6-week course pulmonary rehabilitation.
  Other Names: comparison of d-cycloserine or placebo on enhancing the beneficial effects of pulmonary rehabilitation on breathlessness perception
  Arms: D-cycloserine
Drug: placebo — Other Names:
  comparison of d-cycloserine or placebo on enhancing the beneficial effects of pulmonary rehabilitation on breathlessness perception
  250mg d-cycloserine or identical placebo given immediately to the first 4 sessions of a 6-week course pulmonary rehabilitation
  Other Names: Placebo - identically matched to d-cycloserine containing carrier compound only
  Arms: Drug: d-cycloserine or placebo

SUMMARY:
Dyspnoea is the uncomfortable shortness of breath that debilitates millions of patients with lung disease, heart failure and cancer. It is often very difficult to treat. The sensations of dyspnoea are processed in the brain, and we believe that psychological factors modify and amplify these sensations, frequently exacerbating symptoms.

This study aims to identify the importance of learning in the brain mechanisms of dyspnoea by investigating a cohort of patients with chronic breathlessness undergoing pulmonary rehabilitation . Pulmonary rehabilitation is a six-week course of exercise, education and group therapy that improves dyspnoea but does not improve lung function. This leads us to hypothesise that some of the beneficial effects of PR maybe due to changes in brain processing, potentially relating to a learning effect.

Therefore to probe whether learning is important in the beneficial effects of pulmonary rehabilitation, we intend to modify learning with the drug d-cycloserine. D-cycloserine is an antibiotic that enhances learning due to its effects at N-methyl D-aspartate (NMDA) receptors in the hippocampus. Our previous study in a similar group of patients demonstrated the importance of the hippocampus in breathlessness perception, and we now wish to investigate this in more depth.

The study involves collecting physiological, psychological and clinical measures on in conjunction with brain scanning, before, during and once after pulmonary rehabilitation. Subjects will either receive d-cyloserine or placebo before the first four pulmonary rehabilitation sessions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with chronic lung disease, aged between 45 and 85 years old who have been referred for pulmonary rehabilitation.
* The subject is able and willing to give fully informed consent.

Exclusion Criteria:

Any of the commonly accepted contraindications to MRI scanning, for example, severe claustrophobia, presence of metallic implants, a pacemaker etc.

* Pregnancy. The risk to foetus of radiofrequency energy of the MRI scan is unknown.
* Inadequate understanding of verbal and written information in English, sufficient to complete an MRI safety screening.
* Unable to lie flat and still for 1/2 hour
* Requirements for oxygen therapy
* Significant cardiac, neurological, psychiatric or metabolic disease
* Contra-indications to d-cycloserine: Alcoholism, known hypersensitivity, severe renal failure
* Regular therapy with prescribed opioid analgesics
* Antidepressant therapy (this may alter hippocampal plasticity)
* Previous pulmonary rehabilitation (because the learning may be different on repeat pulmonary rehabilitation treatments)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
BOLD signal changes | baseline, week 3, week 8, 3 months following treatment
  Changes in FMRI BOLD signal in response to breathlessness cues, as a consequence of d-cycloserine administration during pulmonary rehabilitation.

SECONDARY OUTCOMES:
Grey matter volume | baseline, week 3, week 8, 3 months following treatment
  Change in regional brain volume related to changes in breathlessness as a consequence of d-cycloserine administration during pulmonary rehabilitation.

OTHER OUTCOMES:
Grey matter volume compared with healthy controls | baseline, week 3, week 8, 3 months following treatment
  Difference in regional brain volume related to breathlessness in comparison with healthy controls.
difference in BOLD signal compared with healthy controls | baseline, week 3, week 8, 3 months following treatment
  Difference in FMRI BOLD signal in response to breathlessness cues, in comparison with healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle TS Pattinson, BM DPhil FRCA, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Clinical Magnetic Resonance Imaging, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Finnegan SL, Harrison OK, Ezra M, Harmer CJ, Nichols TE, Rahman NM, Reinecke A, Pattinson KTS. The effect of D-cycloserine on brain connectivity over a course of pulmonary rehabilitation - A randomised control trial with neuroimaging endpoints. PLoS One. 2025 Jun 2;20(6):e0323213. doi: 10.1371/journal.pone.0323213. eCollection 2025. PMID 40455920
- [Derived] Finnegan SL, Harrison OK, Booth S, Dennis A, Ezra M, Harmer CJ, Herigstad M, Guillaume B, Nichols TE, Rahman NM, Reinecke A, Renaud O, Pattinson KTS. The effect of d-cycloserine on brain processing of breathlessness over pulmonary rehabilitation: an experimental medicine study. ERJ Open Res. 2023 Apr 3;9(2):00479-2022. doi: 10.1183/23120541.00479-2022. eCollection 2023 Mar. PMID 37020840
- [Derived] Finnegan SL, Browning M, Duff E, Harmer CJ, Reinecke A, Rahman NM, Pattinson KTS. Brain activity measured by functional brain imaging predicts breathlessness improvement during pulmonary rehabilitation. Thorax. 2023 Sep;78(9):852-859. doi: 10.1136/thorax-2022-218754. Epub 2022 Dec 26. PMID 36572534